CLINICAL TRIAL: NCT06159803
Title: LIving BEtteR With asThma - Intervention Development Study
Acronym: LIBERTY-ID
Status: Recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHM MED2028
Record Dates: First submitted 2023-10-17; First posted 2023-12-07 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Adult patients with difficult asthma:
  1. To carry out semi-structured interviews with PDA to explore their experiences, beliefs and attitudes to exercise, diet and emotional self-management support.
  2. To carry out semi-structured interviews with PDA that explores the barriers and facilitators to key behaviours that will be targeted in the intervention.
  3. To carry out iterative think aloud with PDA to elicit feedback on drafts of the intervention to optimise the intervention.
  Interventions: Behavioral: Qualitative Interview
- NHS professionals/Exercise professionals: NHS professionals working with people living with difficult asthma:
  Exercise professionals working with people living with difficult asthma:
  1. To carry out semi-structured interviews with health care and exercise professionals who work with patients living with severe asthma to explore their experiences, beliefs and attitudes to providing exercise, diet and emotional self-management support to this patient group
  2. To carry out semi-structured interviews with health care and exercise professionals who work with patients living with severe asthma that explores the barriers and facilitators to key components that are planned to be included in the intervention.
  3. To carry out iterative think aloud with health care and exercise professionals who work with patients living with severe asthma to elicit feedback on drafts of the intervention to optimise the intervention
  Interventions: Behavioral: Qualitative Interview

INTERVENTIONS:
Behavioral: Qualitative Interview — One-to-one semi-structured interviews and Think Aloud interviews

SUMMARY:
Approximately 330 million people in the world are living with asthma and 3-10% of them has difficult asthma that is challenging to control even with maximum doses of pharmacological treatment. In the last five years our multidisciplinary team has shown the clinical benefits of a short-term structured exercise programme for people living with difficult asthma (PDA) (1). However, engaging PDA in self-maintained exercise long-term and outside of the hospital environment remains a challenge. Changing and maintaining behaviours requires complex psychological and cognitive processes and appropriate modes of support by skilled practitioners. Underpinned by behavioural science and health psychology principles, our team has developed a world renown multimodal self-management support intervention for people living with cancer (2). The intervention focuses on initiating and maintaining exercise, optimising diet and includes supporting people through the cognitive and psychological processes to change their behaviour. We aim to adapt this intervention for PDA to optimise their self-management via the LIBERTY study. To achieve the best outcomes, prior to commencing the LIBERTY study, we aim to develop the intervention using the acclaimed Person-Based Approach (PBA) (3). This methodology is considered gold standard in behaviour change intervention development, implementation and evaluation and maximise the probability of the uptake and maintenance of the desired behaviour.

DETAILED DESCRIPTION:
The burden of poor asthma control remains high in the United Kingdom (UK). Given high asthma prevalence, poor asthma control exerts significant impact at individual and societal levels and accounts for one fifth of the total chronic respiratory disability-adjusted life year burden (4). 'Remission' or well-controlled asthma requires continuation of regular medical treatment, sustained adherence to medications and other self-management behaviours (e.g. healthy diet, avoiding triggers, physical activity), and exposure to risk of potential medication side effects with plus ongoing financial implications. 3-10% of people living with asthma has difficult asthma, defined as asthma that is uncontrolled despite GINA (Global Initiative for Asthma) Step 4 or 5 treatment (5) or requires such treatment to maintain good control and reduce exacerbations. It is increasingly recognised that problematic difficult asthma is a multidimensional state comprising numerous treatable traits that merit targeted approaches (6). This multimorbid disease framework (defined as the coexistence of >2 health conditions) is particularly prevalent in difficult asthma and represents a complex constellation of conditions that collectively impose a significant burden on the patient (7) These treatable traits can be pulmonary, extrapulmonary and behavioural (7). Treatable traits, including obesity, anxiety and depression, dysfunctional breathing and inactivity predict future exacerbation risk in difficult asthma, and so addressing these should be a key part of asthma management for both individual patient benefit and health economic reasons (8). Multimodal non-pharmacological approaches are needed to do that but there is limited understanding of their role in difficult asthma to guide their use.

ELIGIBILITY:
Inclusion Criteria Patient arm:

* Age 18 or over
* Must have had a diagnosis of difficult asthma
* Giving informed consent

Inclusion Criteria Professionals arm:

Aged 18 or over

* Healthcare professional or exercise professional with experience of working with people living
* with difficult asthma
* Giving informed consent

Exclusion Criteria Patient arm:

* Less than 18 years old
* Does not have a diagnosis of difficult asthma
* Unwilling or unable to give informed consent
* Unwilling or unable to participate in the interview
* Participation in the LIBERTY pilot study

Exclusion Criteria Professionals arm:

* Less than 18 years old
* Not a healthcare professional or exercise professional
* Not having experience of working with people living with difficult asthma
* Unwilling or unable to give informed consent
* Unwilling or unable to participate in the interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research population of interest for this study is people living with difficult asthma and health care and exercise professionals working with people with difficult asthma.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-19 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative interviews | 24 months
  Experiences, preferences and perceived barriers to support for exercise, diet and emotional self-management of people living with asthma and professionals working with people living with asthma

CONTACTS AND LOCATIONS:
Locations (1):
- Judit Varkonyi-Sepp, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freeman A, Cellura D, Minnion M, Fernandez BO, Spalluto CM, Levett D, Bates A, Wallis T, Watson A, Jack S, Staples KJ, Grocott MPW, Feelisch M, Wilkinson TMA. Exercise Training Induces a Shift in Extracellular Redox Status with Alterations in the Pulmonary and Systemic Redox Landscape in Asthma. Antioxidants (Basel). 2021 Nov 30;10(12):1926. doi: 10.3390/antiox10121926. PMID 34943027
- [Background] Grimmett C, Bates A, West M, Leggett S, Varkonyi-Sepp J, Campbell A, Davis J, Wootton S, Shaw C, Barlow R, Ashcroft J, Scott A, Moyes H, Hawkins L, Levett DZH, Williams F, Grocott MPW, Jack S. SafeFit Trial: virtual clinics to deliver a multimodal intervention to improve psychological and physical well-being in people with cancer. Protocol of a COVID-19 targeted non-randomised phase III trial. BMJ Open. 2021 Aug 26;11(8):e048175. doi: 10.1136/bmjopen-2020-048175. PMID 34446487
- [Background] Yardley L, Morrison L, Bradbury K, Muller I. The person-based approach to intervention development: application to digital health-related behavior change interventions. J Med Internet Res. 2015 Jan 30;17(1):e30. doi: 10.2196/jmir.4055. PMID 25639757
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] Tay TR, Hew M. Comorbid "treatable traits" in difficult asthma: Current evidence and clinical evaluation. Allergy. 2018 Jul;73(7):1369-1382. doi: 10.1111/all.13370. Epub 2017 Dec 15. PMID 29178130
- [Background] McDonald VM, Hiles SA, Godbout K, Harvey ES, Marks GB, Hew M, Peters M, Bardin PG, Reynolds PN, Upham JW, Baraket M, Bhikoo Z, Bowden J, Brockway B, Chung LP, Cochrane B, Foxley G, Garrett J, Jayaram L, Jenkins C, Katelaris C, Katsoulotos G, Koh MS, Kritikos V, Lambert M, Langton D, Lara Rivero A, Middleton PG, Nanguzgambo A, Radhakrishna N, Reddel H, Rimmer J, Southcott AM, Sutherland M, Thien F, Wark PAB, Yang IA, Yap E, Gibson PG. Treatable traits can be identified in a severe asthma registry and predict future exacerbations. Respirology. 2019 Jan;24(1):37-47. doi: 10.1111/resp.13389. Epub 2018 Sep 19. PMID 30230137
- [Background] Hansen ESH, Pitzner-Fabricius A, Toennesen LL, Rasmusen HK, Hostrup M, Hellsten Y, Backer V, Henriksen M. Effect of aerobic exercise training on asthma in adults: a systematic review and meta-analysis. Eur Respir J. 2020 Jul 30;56(1):2000146. doi: 10.1183/13993003.00146-2020. Print 2020 Jul. PMID 32350100
- [Background] Freitas PD, Ferreira PG, Silva AG, Stelmach R, Carvalho-Pinto RM, Fernandes FL, Mancini MC, Sato MN, Martins MA, Carvalho CR. The Role of Exercise in a Weight-Loss Program on Clinical Control in Obese Adults with Asthma. A Randomized Controlled Trial. Am J Respir Crit Care Med. 2017 Jan 1;195(1):32-42. doi: 10.1164/rccm.201603-0446OC. PMID 27744739
- [Background] Paolucci EM, Loukov D, Bowdish DME, Heisz JJ. Exercise reduces depression and inflammation but intensity matters. Biol Psychol. 2018 Mar;133:79-84. doi: 10.1016/j.biopsycho.2018.01.015. Epub 2018 Feb 3. PMID 29408464
- [Background] Cordova-Rivera L, Gibson PG, Gardiner PA, McDonald VM. A Systematic Review of Associations of Physical Activity and Sedentary Time with Asthma Outcomes. J Allergy Clin Immunol Pract. 2018 Nov-Dec;6(6):1968-1981.e2. doi: 10.1016/j.jaip.2018.02.027. Epub 2018 Mar 3. PMID 29510231
- [Background] Garcia-Aymerich J, Varraso R, Anto JM, Camargo CA Jr. Prospective study of physical activity and risk of asthma exacerbations in older women. Am J Respir Crit Care Med. 2009 Jun 1;179(11):999-1003. doi: 10.1164/rccm.200812-1929OC. Epub 2009 Feb 26. PMID 19246716
- [Background] Freeman AT, Hill D, Newell C, Moyses H, Azim A, Knight D, Presland L, Harvey M, Haitchi HM, Watson A, Staples KJ, Kurukulaaratchy RJ, Wilkinson TMA. Patient perceived barriers to exercise and their clinical associations in difficult asthma. Asthma Res Pract. 2020 Jun 9;6:5. doi: 10.1186/s40733-020-00058-6. eCollection 2020. PMID 32537235
- [Background] Azim A, Freeman A, Lavenu A, Mistry H, Haitchi HM, Newell C, Cheng Y, Thirlwall Y, Harvey M, Barber C, Pontoppidan K, Dennison P, Arshad SH, Djukanovic R, Howarth P, Kurukulaaratchy RJ. New Perspectives on Difficult Asthma; Sex and Age of Asthma-Onset Based Phenotypes. J Allergy Clin Immunol Pract. 2020 Nov-Dec;8(10):3396-3406.e4. doi: 10.1016/j.jaip.2020.05.053. Epub 2020 Jun 13. PMID 32544545
- [Background] Varkonyi-Sepp J, Freeman A, Ainsworth B, Kadalayil LP, Haitchi HM, Kurukulaaratchy RJ. Multimorbidity in Difficult Asthma: The Need for Personalised and Non-Pharmacological Approaches to Address a Difficult Breathing Syndrome. J Pers Med. 2022 Aug 31;12(9):1435. doi: 10.3390/jpm12091435. PMID 36143220
- [Background] Morrison L, Muller I, Yardley L, Bradbury K. The person-based approach to planning, optimising, evaluating and implementing behavioural health interventions. The European Health Psychologist. 2018;20(3):464-9
- [Background] Bourgeault, I., Dingwall, R., & De Vries, R. (Eds.). (2010). The SAGE handbook of qualitative methods in health research. Sage Publications Ltd., London
- See also: Asthma GIf. Global Strategy for Asthma Management and Prevention 2021 — https://ginasthma.org/wp-content/uploads/2021/05/GINA-Main-Report-2021-V2-WMS.pdf.
- See also: Braun V, Clarke V. Using thematic analysis in psychology Using thematic analysis in psychology. Qual Res Psychol [Internet]. 206AD;3:77-101 — http://www.ncbi.nlm.nih.gov/pubmed/11752478
- See also: HRA guidance — http://www.hra.nhs.uk/resources/after-you-apply/amendments/
- See also: ICMJE - Roles and Responsibilities of Authors, Contributors, Reviewers, Editors, Publishers, and Owners — https://www.icmje.org/recommendations/browse/roles-and-responsibilities/defining-the-role-of-authors-and-contributors.html